CLINICAL TRIAL: NCT00281606
Title: A Phase IV, Randomized, Open-label Study of the Tolerability of Once Daily Lopinavir/Ritonavir (LPV/r) Liquid Versus Capsules
Brief Title: A Multicenter Study to Assess the Tolerability of Once Daily Lopinavir/Ritonavir (LPV/r) Liquid Versus Capsules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, J Allen McCutchan, Prof Emeritus, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCTG 585
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: HIV Infection
Keywords: Lopinavir; antiretroviral therapy; cross-over; tolerability
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Lopinavir

ARMS (2):
- LPV/r (800/200 mg) 10 ml liquid (Active Comparator): Once daily Lopinovir/ritonavir (800/200 mg) taken as a 10 ml liquid
  Interventions: Drug: Different formulations of once-daily lopinavir/ritonavir
- LPV/r (800/200 mg) 6 gel capsules (Active Comparator): Once daily Lopinavir/ritonavir (800/200 mg) as 6 gel capsules
  Interventions: Drug: Different formulations of once-daily lopinavir/ritonavir

INTERVENTIONS:
Drug: Different formulations of once-daily lopinavir/ritonavir — CCTG585 is a randomized, open-label, two arm cross-over study to compare the tolerability of once daily LPV/r liquid versus capsules
  Other Names: Lopinavir/Ritonavir (LPV/r)

SUMMARY:
Guidelines have continued to list lopinavir/ritonavir as a preferred protease inhibitor-containing regimen for HIV-infected individuals. There has recently been increasing interest in once daily therapy. While lopinavir/ritonavir has recently been approved as a once daily therapy it was associated with considerable diarrhea in those treated with soft gel capsules. It is the hope that alternative formulations of lopinavir/ritonavir may provide similar pharmacokinetics with improved tolerability. This includes the possibility of using liquid or newly released tablets. This study will treat people tolerating their current regimen with up to four weeks of each formulation with several assessments of pharmacokinetics and tolerability for each.

DETAILED DESCRIPTION:
This study is designed to assess the tolerability of different forms (liquid, capsules or tablets) of lopinavir/ritonavir given once-daily as part of combination therapy for HIV infection. Study subjects will be those tolerating a stable regimen of HIV medications with undetectable levels of HIV in their blood. They will be assigned by chance to receive once daily liquid or soft gel capsules of lopinavir/ritonavir for up to four weeks. At that time they will receive the alternative formulation for up to four weeks. They will then be given once daily lopinavir/ritonavir in the recently released tablet formulation. After up to four weeks of each of these formulations several assessments will be made of the overall tolerability of the drug. After four weeks of tablets they will be allowed to take whatever regimen they want and will be followed for an additional 36 weeks for a total duration of study of up to 48 weeks. The pharmacokinetics of each formulation of lopinavir/ritonavir given once daily will also be assessed in a subset of study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness of subject or legal guardian/representative to give written informed consent.
* HIV-1 infected.
* At least 18 years of age
* Have the last two HIV-1 RNA measurements performed prior to screening be <50 or 75 copies/mL within the last 180 days, as well as at the time of screening.
* No evidence of primary PI mutations (defined by IAS-USA) documented on previous resistance testing, if ever performed and available, or suggested to be present by previous treatment history.
* Laboratory values:

  * Absolute neutrophil count (ANC) >500/mm3.
* -Hemoglobin >7.0 g/dL.

  * platelet count >50,000/mm3.
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase <5 X ULN.
  * Total bilirubin <2.5 x ULN, unless on IDV or ATV in which case must be <1.5 x ULN of direct bilirubin.
  * Calculated creatinine clearance >50 mL/min as estimated by the Cockcroft-Gault equation
* For women of reproductive potential, negative serum or urine pregnancy test within 7 days prior to initiating study medications. If participating in sexual activity that could lead to pregnancy, female study subjects must use two forms of contraception, one of which must be a barrier method. All subjects must continue to use contraception for 6 weeks after stopping the study medications.
* Willingness to take an alcohol containing product.
* Karnofsky performance score >70.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Greater than Grade 1 diarrhea or nausea (as defined by protocol)
* Use of a NNRTI within 12 weeks of screening
* Use of antimotility or antiemetics during the 14 days prior to screening
* Use of any of the prohibited medications (defined by protocol) within 30 days of study entry.
* Need to continue the use of prohibited or select precautionary medications (defined by protocol)
* Known hypersensitivity to lopinavir/ritonavir
* Active drug or alcohol use or dependence which, in the Investigator's opinion, may interfere with adherence to study requirements or endanger subject's health while on the study
* Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 30 days prior to study entry.
* Acute therapy for serious infection or other serious medical illnesses (in the judgment of the site investigator) requiring systemic treatment and/or hospitalization within 14 days prior to study entry.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV-1 vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-02-14 (Actual); Primary Completion 2007-10-16 (Actual); Study Completion 2012-06-13 (Actual)

PRIMARY OUTCOMES:
Measuring whether the subject has severity of diarrhea grade 2 or higher or exhibits treatment-limiting toxicity when treated with once daily Lopinavir/ritonavir [LPV/r] (800/200 mg) as 10 ml liquid vs. 6 soft gel capsules. | Baseline to week 48
  To assess the comparative tolerability of once daily Lopinavir/ritonavir [LPV/r] (800/200 mg) as 10 ml liquid vs. 6 soft gel capsules by measuring incidence rates as assessed by the CTCAE v4.0 in each arm of: a) grade 2 or higher diarrhea plus b) dose limiting toxicity of any kind.

SECONDARY OUTCOMES:
Incidence Measures of Treatment-limiting toxicity | Baseline to week 48
  Separately evaluating at the end of week 4 or at the time therapy is discontinued for treatment-limiting toxicity of the two 4 week phases of the cross-over trial (Steps 1 and 2).
Incidence Measures of Drug-related diarrhea | Baseline to week 48
  Separately evaluating at the end of week 4 or at the time therapy is discontinued for drug-related diarrhea of the two 4 week phases of the cross-over trial (Steps 1 and 2).
Incidence Measures of the Use of antiemetic and/or antimotility therapy | Baseline to week 48
  Separately evaluating at the end of week 4 or at the time therapy is discontinued for antiemetic and/or antimotility therapy of the two 4 week phases of the cross-over trial (Steps 1 and 2).
Incidence Measures of Adverse events other than nausea and diarrhea | Baseline to week 48
  Separately evaluating at the end of week 4 or at the time therapy is discontinued for adverse events other than nausea and diarrhea of the two 4 week phases of the cross-over trial (Steps 1 and 2).
Incidence Measures of Laboratory abnormalities, e.g. lipids, liver enzymes | Baseline to week 48
  Separately evaluating at the end of week 4 or at the time therapy is discontinued for laboratory abnormalities of the two 4 week phases of the cross-over trial (Steps 1 and 2).
Incidence Measures of HIV RNA suppression to <50 copies/ml | Baseline to week 48
  Separately evaluating at the end of week 4 or at the time therapy is discontinued for HIV RNA suppression to <50 copies/ml of the two 4 week phases of the cross-over trial (Steps 1 and 2).
Preference for Lopinavir/ritonavir liquid, capsules or tablets, and the degree of like or dislike of each | Week 8 and week 48
  The stated preference for LPV/r liquid, capsules or tablets, and the degree of like or dislike of each in those who choose an option other than once daily LPV/r tablets at start of Step 4
Evaluating the proportion of screened individuals who choose not to be randomized after the liquid Lopinavir/ritonavir taste test | Baseline
  Evaluating the proportion of screened individuals who choose not to be randomized after the liquid LPV/r taste test at the time of enrollment into the study
Evaluating the severity of diarrhea | Week 4, week 8 and week 48
  Measuring sum of days with diarrhea weighted for highest level of severity (sum of event severity numbers = 1-5) on that day via the Division of AIDS Table for Grading Adult Adverse Experiences that can be found on the ROC Web site: http://rcc.tech-res-intl.com/
Evaluating the severity of nausea | Week 4, week 8 and week 48
  Measuring days of nausea weighted for the highest level of severity (sum of event severity numbers = 1-5) on that day via the Division of AIDS Table for Grading Adult Adverse Experiences that can be found on the ROC Web site: http://rcc.tech-res-intl.com/
Evaluating proportion with plasma HIV RNA <50 copies/mL at the end of Step 4 | Week 4, week 8 and week 48
  Evaluating the proportion of participants with plasma HIV RNA <50 copies/mL at the end of Step 4

OTHER OUTCOMES:
Direct inspection of Pre-dose concentrations (Cpre-dose) for Lopinavir/ritonavir (LPV/r) | Baseline and 12 weeks
  Direct inspection of the concentration data to assess Pre-dose concentrations (Cpre-dose) for Lopinavir/ritonavir (LPV/r) liquid, capsules and tablets
Direct inspection of trough concentrations (Ctrough) for Lopinavir/ritonavir (LPV/r) | Baseline and 12 weeks
  The magnitude of difference within patients of the two formulations will be assessed with the Wilcoxon signed-rank test. The trough concentrations of the Group 2 subjects may also be compared using the Wilcoxon signed-rank test to detect a difference between the formulations.
Direct inspection of 24-hour post-dose concentrations (C24) for Lopinavir/ritonavir (LPV/r) | Baseline and 12 weeks
  Model dependent and independent traditional pharmacokinetic approaches will be used to estimate pharmacokinetic parameters, such as the area under the concentration versus time curve from time 0 to 24 hours (AUC0-24).
Direct inspection of maximum plasma concentrations (Cmax) for Lopinavir/ritonavir (LPV/r) | Baseline and 12 weeks
  Determine TDF plasma and urine concentrations in Group 1 patients taking TDF concurrently with LPV/r (Group 3).
Direct inspection of the corresponding time to Cmax (Tmax) for Lopinavir/ritonavir (LPV/r) | Baseline and 12 weeks
  Model dependent and independent traditional pharmacokinetic approaches will be used to estimate pharmacokinetic parameters, such as the area under the concentration versus time curve from time 0 to 24 hours (AUC0-24), the terminal half-life (t1/2), the apparent clearance (CL/F), and the apparent volume of distribution (Vz/F).
Estimation of concentration versus time curve from time 0 to 24 hours (AUC0-24) for Lopinavir/ritonavir (LPV/r) | Baseline and 12 weeks
  Model dependent and independent traditional pharmacokinetic approaches will be used to estimate concentration versus time curve from time 0 to 24 hours (AUC0-24). The AUC0-24 and Cmax ratios of liquid to capsule LPV/r within subjects will be used to assess bioequivalence.
Estimation of terminal half-life (t1/2) for Lopinavir/ritonavir (LPV/r) | Baseline and 12 weeks
  Model dependent and independent traditional pharmacokinetic approaches will be used to estimate terminal half-life (t1/2)
Estimation of apparent clearance (CL/F) for Lopinavir/ritonavir (LPV/r) | Baseline and 12 weeks
  Model dependent and independent traditional pharmacokinetic approaches will be used to estimate apparent clearance (CL/F)
Estimation of apparent volume of distribution (Vz/F) for Lopinavir/ritonavir (LPV/r) | Baseline and 12 weeks
  Model dependent and independent traditional pharmacokinetic approaches will be used to estimate apparent volume of distribution (Vz/F)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Daar, MD, Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - UCI, Irvine, California
  - USC, Los Angeles, California
  - UCSD, San Diego, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Harbor-UCLA Medical Center, Torrance, California

REFERENCES:
- [Result] 1. Best B, Rieg G, Sun S, Jain S, Kemper C, Diamond C, Hermes A, Haubrich R, Daar E, and California Collaborative Treatment Group (CCTG) 585 Team. Increased lopinavir concentrations on once-daily tablets as compared with capsules and liquid formulations. 15th Conference on Retroviruses and Opportunistic Infections; February 3-6, 2008; Boston, MA. Abstract 766a. 2. CDB088 Abstract Switching to once-daily (QD) lopinavir/ritonavir (LPV/r) liquid (Liq), capsules (caps) and tablets (tabs): a randomized, ppen label, cross-over study (CCTG 585). 5th IAS Conference on HIV Pathogenesis, Treatment and Prevention; Cape Town 2009 G. Rieg1, S. Jain2, S. Sun2, R. Larsen3, C. Kemper4, C. Diamond5, S. Schneider6, D. Shamblaw7, A. Hermes8, R. Haubrich9, E. Daar10, California Collaborative Treatment Group (CCTG)